CLINICAL TRIAL: NCT03966261
Title: INcrétines et REModelage OSseux
Brief Title: The Role of Incretins in Bone Remodeling in Humans
Acronym: INCREMOS
Status: Terminated | Type: Observational
Why Stopped: No more inclusion needed for primary critera analysis
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-A01632-53
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Incretins; Osteoporosis; Bone Remodeling; Healthy
MeSH Terms: conditions — Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample — we perform blood sample in healthy subject before and after a meal to measure incretins concentration

SUMMARY:
The role of incretins (GIP and GLP-1) on cells and bone tissue has been shown in cellular and animal studies. In humans, the role of these hormones is mainly studied in the pathophysiology of diabetes, their effect on bone is unknown. The serum incretin concentration is low and increases rapidly after a meal. This increase is brief, incretins being rapidly degraded by dipeptidylpeptidase 4 (DPP-4). The dosage of these hormones is complex and the basal "normal" serum concentrations and after feeding in healthy subjects are unknown. Before any study on the effect of incretins on bone remodeling in humans, it is necessary to establish physiological concentrations of incretins in healthy subjects.

The aim of this study is to estimate physiological concentrations of incretins in healthy subject.

ELIGIBILITY:
Inclusion Criteria:

* healthy women and men

Exclusion Criteria:

* known osteoporosis
* osteoporotic fracture
* tobacco
* alcohol : > 2 glasses/day
* type 1 and type 2 diabetes
* BMI < 19kg/m² or > 30kg/m²
* heart failure, kidney failure
* cancer
* bariatric surgery
* graft
* cirrhosis
* use in the past year : bisphosphonate, denosumab, raloxifene, teriparatide, oral or IV glucocorticoid during 3 months or more

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and men aged from 30 to 70 years without bone patholog nor pathological condition influencing bone remodeling nor treatment influencing bone remodeling
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
incretins concentrations before and after a meal in healthy subjects | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mabilleau G. Interplay between bone and incretin hormones: A review. Morphologie. 2017 Mar;101(332):9-18. doi: 10.1016/j.morpho.2016.06.004. Epub 2016 Aug 8. PMID 27423214
- [Background] Mabilleau G, Gobron B, Mieczkowska A, Perrot R, Chappard D. Efficacy of targeting bone-specific GIP receptor in ovariectomy-induced bone loss. J Endocrinol. 2018 Nov;239(2):215-227. doi: 10.1530/JOE-18-0214. PMID 30121578
- [Background] Mabilleau G, Gobron B, Bouvard B, Chappard D. Incretin-based therapy for the treatment of bone fragility in diabetes mellitus. Peptides. 2018 Feb;100:108-113. doi: 10.1016/j.peptides.2017.12.008. PMID 29412811